CLINICAL TRIAL: NCT00917189
Title: Computer-Based Cognitive Remediation in Adolescents With VCFS
Brief Title: Computerized Cognitive Skills Training for Adolescents With Velocardiofacial Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R33MH085901 (NIH); R33MH085901 (NIH); DDTR B4-TBI
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Velocardiofacial Syndrome
Keywords: VCFS; Chromosome 22q Deletion Syndrome; Learning Disorders
MeSH Terms: conditions — DiGeorge Syndrome; Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Computerized Cognitive Skills Training (Experimental): Participants will receive the Challenging Our Minds intervention, delivered in-person in Phase 1 and remotely in Phases 2 and 3.
  Interventions: Behavioral: Challenging Our Minds Program

INTERVENTIONS:
Behavioral: Challenging Our Minds Program — A computerized cognitive intervention that provides training in attention, memory, and executive function

SUMMARY:
This study will test a computer-based treatment for youth with the genetic disorder velocardiofacial syndrome (VCFS) to help them improve skills in memory, attention, and executive functioning.

DETAILED DESCRIPTION:
Velocardiofacial syndrome (VCFS) is a genetic condition caused by deletion of a segment of the 22nd chromosome at the location 22q11.2. VCFS is characterized by a combination of medical problems related to the palate (velo) and the heart (cardio) and by a distinct facial appearance. Also common in people with VCFS, among other problems, are learning and speech difficulties. These difficulties are specifically categorized as deficits in attention, working memory, and executive functioning. This study will develop and test a computer-based intervention for adolescents with VCFS that will teach them cognitive skills to lessen these deficits.

This study will have three phases. In the first phase, the intervention will be pilot tested with an in-person coach. In the second phase, the intervention will be pilot tested remotely with a video-conferencing coach. In the third phase, the intervention will be delivered remotely, and testing will be expanded to include more participants and a longer assessment period. Information on participant drop-out and level of difficulty will be gathered and used to refine the treatment between phases.

Participation in Phase 1 will last 6 months. At study entry, participants will complete baseline measures that involve a structured diagnostic interview to assess behavioral or emotional difficulties and cognitive testing to assess intellectual functioning. Then they will meet with a study training coach three times a week at their homes. During these sessions, participants will complete exercises in the Challenging our Minds program, a computer-based system designed to improve learning. Exercises will develop skills in seven domains: attention, decision making, memory, understanding relationships between objects, problem solving, communication, and social perception.

Participation in Phase 2 will last 6 to 9 months. Participants in this phase will complete the same baseline measures that occurred at study entry and then complete exercises in Challenging our Minds three times a week. Instead of having a training coach come to their homes, participants in Phase 2 will work with a training coach via video-conferencing software.

Participation in Phase 3 will last 2 years. Participants will undergo assessments at four points: at baseline, after 9 months, after 18 months, and after 27 months. These assessments will include the baseline measures from the previous phases as well as a virtual reality computer task. Between their visits at 9 and 18 months, participants will work with a training coach via video conferencing three times a week to complete the Challenging our Minds exercises.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of velocardiofacial syndrome (VCFS)
* IQ score between 70 and 90

Exclusion Criteria:

* Presence of psychotic symptoms

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2009-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The California Learning Test and the Visual Span Test | Measured immediately following the intervention at each phase

SECONDARY OUTCOMES:
Performance on the Apartment Test | Measured immediately following the intervention at each phase

CONTACTS AND LOCATIONS:
Overall Officials: Wendy R. Kates, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Result] Mariano MA, Tang K, Kurtz M, Kates WR. Examining the durability of a hybrid, remote and computer-based cognitive remediation intervention for adolescents with 22q11.2 deletion syndrome. Early Interv Psychiatry. 2018 Aug;12(4):686-693. doi: 10.1111/eip.12367. Epub 2016 Sep 15. PMID 27629273
- [Result] Mariano MA, Tang K, Kurtz M, Kates WR. Cognitive remediation for adolescents with 22q11 deletion syndrome (22q11DS): a preliminary study examining effectiveness, feasibility, and fidelity of a hybrid strategy, remote and computer-based intervention. Schizophr Res. 2015 Aug;166(1-3):283-9. doi: 10.1016/j.schres.2015.05.030. Epub 2015 Jun 1. PMID 26044111